CLINICAL TRIAL: NCT02130115
Title: LungPoint ATV for Biopsy in Patients Undergoing Lobectomy
Acronym: LABEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Broncus Medical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Protocol 40
Record Dates: First submitted 2014-04-25; First posted 2014-05-05 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: LungPoint ATV System — The LungPoint ATV System is an image-guided navigation system used to access tissue samples in the lungs.

SUMMARY:
The purpose of this study is to evaluate the safety and performance of the LungPoint ATV System.

DETAILED DESCRIPTION:
The LungPoint ATV System is an image-guided navigation system used to access tissue samples in the lungs. This feasibility study is being conducted to assess the ability of the investigator to access and sample tissue using this system in patients undergoing lobectomy or pneumonectomy. Navigation to and sampling of the patient's lung cancer tumor is conducted immediately prior to the scheduled lobectomy or pneumonectomy.

Note: This study was conducted as a single-center feasibility clinical trial to determine the feasibility of this device. The primary outcome measures related only to feasibility and not to health outcomes. Therefore it was not registered on clinicaltrials.gov prior to the start of enrollment. Subsequently, it was determined that the results were compelling and therefore it was registered to facilitate publication.

ELIGIBILITY:
Inclusion Criteria:

1. Surgical candidates age 21-75 years at screening
2. Known or suspected lung cancer or intrapulmonary metastatic disease with SPN greater than 10 mm and less than 40mm in largest dimension
3. No known endobronchial tumor
4. Tumor located anywhere in parenchymal tissue >1 cm from pleura and accessible bronchoscopically through a POE.
5. Willing to participate in all aspects of study protocol for duration of study
6. Able to understand study requirements
7. Signs study-related informed consent document

Exclusion Criteria:

1. Any contraindication to bronchoscopy, for example: (a.) Untreatable life-threatening arrhythmias, (b.) Inability to adequately oxygenate the patient during the procedure, (c.) Acute respiratory failure with hypercapnia (unless the patient is intubated and ventilated), (d.) Recent myocardial infarction, (e.) Previously diagnosed high-grade tracheal obstruction, (f.) Uncorrectable coagulopathy.
2. Known coagulopathy
3. Platelet dysfunction or platelet count < 100 x 103 cells/mm3
4. History of major bleeding with bronchoscopy
5. Pulmonary hypertension with mean PAP >25 mm
6. Moderate-to-severe pulmonary fibrosis
7. Moderate to severe emphysema or COPD with FEV1 <60% predicted or RV >200% predicted
8. Bullae >5 cm located in vicinity of target SPN or ATV tunnel
9. Any other severe or life-threatening comorbidity that could increase the risk of bronchoscopic biopsy or ATV tunneling, for example: (a.) ASA class > 3, (b.) > stage 3 heart failure, (c.) severe cachexia, (d.) severe respiratory insufficiency or hypoxia
10. Ongoing systemic infection
11. Contraindication to general anesthesia
12. Chronic use of anticoagulants (e.g., heparin, Warfarin) or antiplatelet agents (e.g. aspirin, clopidogrel)
13. Participation in any other study in last 30 days
14. Prior thoracic surgery on the same side of the lung as the SPN
15. Breastfeeding women or females of childbearing potential with a positive pregnancy test prior to the procedure or the intent to become pregnant during the study.
16. Life expectancy of less than one year.
17. Patients with known intrapulmonary metastases of extrapulmonary cancer/tumors

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Ability to complete procedure using system | At completion of procedure
  The proportion of cases (attempted nodules) in which the procedure could be substantially completed by the investigator divided by the number of cases (nodules) for which at least one attempt to pass any LungPoint study device into the bronchoscope was made.

SECONDARY OUTCOMES:
Proportion of nodules biopsied yielding tissue sufficient for diagnosis | Upon asssessment of histology of tissue sample taken during procedure
  The number of nodules with at least one biopsy sufficient for a tissue diagnosis divided by the number of nodules sampled using the LungPoint ATV system.
Number of significant adverse events | Up through lobectomy of lobe at end of procedure
  The number of SAEs rated as probably or definitely related to the study device and/or procedure divided by the number of patients in whom an attempt at study device use was made. The adverse events specifically tracked in this study are hemoptysis and pneumothorax.

CONTACTS AND LOCATIONS:
Overall Officials: Felix Herth, MD, Principal Investigator — Heidelberg University
Locations (1):
- Thoraxklinik, Heidelberg, Germany

REFERENCES:
- [Derived] Herth FJ, Eberhardt R, Sterman D, Silvestri GA, Hoffmann H, Shah PL. Bronchoscopic transparenchymal nodule access (BTPNA): first in human trial of a novel procedure for sampling solitary pulmonary nodules. Thorax. 2015 Apr;70(4):326-32. doi: 10.1136/thoraxjnl-2014-206211. Epub 2015 Mar 6. PMID 25746631